CLINICAL TRIAL: NCT07261956
Title: Usefulness of Lung Ultrasound for the Detection of Volume Overload in Patients With Severe Preeclampsia
Brief Title: Lung Ultrasound for the Detection of Volume Overload in Patients With Severe Preeclampsia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Head of Research Department, Saint Thomas Hospital, Panama
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4377
Record Dates: First submitted 2025-08-24; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Edema - Acute; Preeclampsia
Keywords: Pulmonary edema; Severe preeclampsia; B lines; Lung ultrasound
MeSH Terms: conditions — Pre-Eclampsia; Pulmonary Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Severe preeclampsia (Experimental): Pregnant subjects (24 weeks - 41 weeks) with severe preeclampsia
  Interventions: Diagnostic Test: Lung ultrasound

INTERVENTIONS:
Diagnostic Test: Lung ultrasound — Lung ultrasounf at three moments (at admission, before delivery and immediate post partum) to determine B Lines

SUMMARY:
This research aims to evaluate the usefulness of lung ultrasound (LUS) for detecting and monitoring fluid overload in patients with severe preeclampsia. Severe preeclampsia is a leading cause of maternal death and illness worldwide, often causing fluid buildup that can lead to a serious complication called pulmonary edema, especially after delivery.

The study will be a prospective, longitudinal observational study with a diagnostic validation component. It will involve patients with a diagnosis of severe preeclampsia who meet specific inclusion criteria. Each participant will undergo a clinical exam and a lung ultrasound, which will assess eight zones of the lungs. The total number of B-lines-a sign of interstitial edema-will be documented.

Data will be collected at three key times: upon admission, in the immediate postpartum period (within 24 hours of delivery), and 7-10 days postpartum. The results from the LUS will be compared to clinical signs like shortness of breath, rapid breathing, crackling sounds in the lungs, and oxygen saturation levels.

The expected impact of this research is to provide evidence that LUS is a valuable, non-invasive, and accessible tool for the early detection of pulmonary congestion in patients with severe preeclampsia. This could lead to improved clinical decision-making and a reduction in maternal respiratory complications.

ELIGIBILITY:
Inclusion Criteria:

* Preeclampsia with severe features.
* Gestational age 24 weeks - 41 weeks.

Exclusion Criteria:

* Chronic lung disease.
* Known heart disease.
* Diagnosis of lung edema at admission
* Body mass index > 40
* Need for immediate delivery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Lung Ultrasound evaluation | One evaluation at admission, another one just before delivery and a final one 24 hours after delivery
  Three or more B Lines in at least two lung zones using lung ultrasound

SECONDARY OUTCOMES:
Dyspnea | Report of the symptom by the patient from admission for up to three days
  Subjective sensation of difficulty breathing
Tachypnea | Report of the symptom from admission for up to three days.
  Respiratory rate above 20 breaths/min
Oxygen saturation | Report of the value measured by a pulse oxymeter from admission for up to three days
  Oxygen saturation measured by pulse oxymeter

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo Reyes, MD, Study Director — Saint Thomas Hospital, Panama
Locations (1):
- Saint Thomas Hospital, Panama City, Provincia de Panamá, Panama

IPD SHARING:
Plan to Share IPD: No